CLINICAL TRIAL: NCT06214117
Title: Comparison of Emergence Agitation in Children Following Tonsillectomy and Adenoidectomy Under Remimazolam or Sevoflurane General Anesthesia
Brief Title: Comparison of Emergence Delirium: Remimazolam vs Sevoflurane Anesthesia
Acronym: CEDCRSA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SAHoWMU-CR2024-03-103
Record Dates: First submitted 2024-01-08; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — remimazolam; Anesthesia, Intravenous; Sevoflurane; Anesthesia, Inhalation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group R (Experimental): Induction of anesthesia:Anesthesia will induced with remimazolam at 0.3-0.5 mg/kg; Maintenance of anaesthesia:Remimazolam will infuse initially at a rate of 2 mg/kg/h (1-3 mg/kg/h).
  Interventions: Drug: Remimazolam
- Group S (Placebo Comparator): Induction of anesthesia:Anesthesia will induced with 8% sevoflurane in 100% oxygen at flow rate of 6 L/min; Maintenance of anaesthesia:Anesthesia depth was maintained at 1-1.5 MAC by sevoflurane.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Remimazolam — Anesthesia induction:intravenous Fentanyl 2-3 μg/kg, remimazolam 0.3-0.5 mg/kg and Rocuronium 0.6mg/kg; Maintenance of anesthesia:Remimazolam will infuse initially at a rate of 2 mg/kg/h (1-3 mg/kg/h), and remifentanil will administer at an initial infusion rate of 0.25 μg/kg/min (0.1-0.5 μg/kg/min).
  Other Names: intravenous anesthesia
  Arms: Group R
Drug: Sevoflurane — Anesthesia induction: Anesthesia will induce with 8% sevoflurane in 100% oxygen at flow rate of 6 L/min, and then intravenous fentanyl (2-3 μg/kg) and rocuronium (0.6 mg/kg); Maintenance of anaesthesia: Anesthesia depth will maintain at 1-1.5 minimum alveolar concentration (MAC), and remifentanil was infuse at an initial rate of 0.25 μg/kg/min (0.1-0.5 μg/kg/min).
  Other Names: inhalation anesthesia
  Arms: Group S

SUMMARY:
Emergence delirium can lead to a range of clinical problems and is even associated with short-term behavioral changes in children. Pediatric ear, nose, and throat (ENT) surgery is one of the most common surgical types for postoperative delirium in children. Sevoflurane anesthesia is also a known cause of postoperative delirium. Therefore, this study aims to explore whether there is a difference in the incidence of postoperative delirium in children under remimazolam general anesthesia and sevoflurane anesthesia.

DETAILED DESCRIPTION:
children aged 3-6 years old were randomly and equally allocated into two groups: Group R remimazolam, Group S with sevoflurane, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-6 years;
2. American Society of Anaesthesiologist (ASA) I or II;
3. Booked for Tonsillectomy and Adenoidectomy;
4. BMI for age between the 25th and 85th percentiles according to the 2000 Centers for Disease Control and Prevention (CDC) growth charts.

Exclusion Criteria:

1. Children (ASA III- IV) who had abnormal liver and kidney function, cardiovascular, endocrine dysfunction, or any other organ dysfunction;
2. Allergy or hypersensitive reaction to remimazolam;
3. mental disorder
4. Recently respiratory infection;
5. Other reasons that researchers hold it is not appropriate to participate in this trial: under specialized care or lived in social welfare institutions, or any other factors that could affect their ability to participate in the study.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
The incidence of emergence delirium | Within up to 30 minutes after operation
  The pediatric anesthesia emergence delirium scale consists of four items. Each item is scored 0-4 yielding a total between 0 and 20.The degree of emergence delirium increased directly with the total score.
  Pediatric anesthesia emergence delirium scale ≥10 at any time indicates presence of emergence delirium.

SECONDARY OUTCOMES:
Pediatric anesthesia emergence delirium | Within up to 30 minutes after operation
  The pediatric anesthesia emergence delirium scale consists of four items. Each item is scored 0-4 yielding a total between 0 and 20.
  The degree of emergence delirium increased directly with the total score.
The Face, Legs, Activity, Cry, Consolability Scale (FLACC) | Within up to 30 minutes after operation
  The FLACC scale consists of five items. Each item is scored 0-2 yielding a total between 0 and 10.
  The degree of pain increased directly with the total score.
Extubation time | Within up to 30 minutes after operation
  The time from discontinuation of anesthesia drug to extubation.
Recovery times | Within up to 30 minutes after operation
  The time from discontinuation of anesthesia drug to the first open eye of the children and to achieve aldrete≥9
PHBQ-AS | 3 days after operation
  Post-Hospitalization Behavior Questionnaire for Ambulatory Surgery (PHBQ-AS) is a parental report measure used to assess negative behavior change after hospitalization, consisting of 11 items on 1-5 score. The PHBQ-AS score will be calculated for each respondent as the mean score of all individual items answered on the questionnaire.
  A score above 3 will indicate the presence of negative behavioral change, a score equal to 3 will indicate no behavioral change, and a score below 3 will indicate an improvement in behavior.
Number of children with adverse effects | Up to 24 hours including intraoperative, and postoperative periods
  Bradycardia and/or hypotension need for hemodynamic support Desaturation is defined as Oxygen desaturation <90% Any adverse effects requiring interventions

CONTACTS AND LOCATIONS:
Overall Officials: Huacheng Liu, Ph.D., Principal Investigator — The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University
Locations (1):
- The second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Ma HY, Cai YH, Zhong JW, Chen J, Wang Z, Lin CY, Wang QQ, Liu HC. The effect of remimazolam-based total intravenous anesthesia versus sevoflurane-based inhalation anesthesia on emergence delirium in children undergoing tonsillectomy and adenoidectomy: study protocol for a prospective randomized controlled trial. Front Pharmacol. 2024 Jun 25;15:1373006. doi: 10.3389/fphar.2024.1373006. eCollection 2024. PMID 38983921